CLINICAL TRIAL: NCT04350216
Title: Effect of Sarilumab Therapy on Atherosclerotic Disease Assessed by Positron Emission Tomography/Computed Tomography (PET/CT) in Patients With Rheumatoid Arthritis
Brief Title: Effect of Sarilumab on Atherosclerotic Disease Assessed by PET/CET in Patients With RA (SARIPET)
Acronym: SARIPET
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Instituto de Investigación Marqués de Valdecilla (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SARIPET_2019.099
Record Dates: First submitted 2020-04-08; First posted 2020-04-16 (Actual); Last update posted 2020-04-27 (Actual); Status verified 2020-04

CONDITIONS: Rheumatoid Arthritis; Atherosclerosis
Keywords: Positron Emission Tomography; chronic inflammatory state; interleukin (IL)-6; Computed Tomography
MeSH Terms: conditions — Arthritis, Rheumatoid; Atherosclerosis | interventions — sarilumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sarilumab therapy (Experimental): Patients will be treated every two weeks with 200 mg of the anti-IL human monoclonal antibody-6Rα Sarilumab (Kevzara) with or without conventional DMARDs. Sarilumab administration will be subcutaneous (abdomen, thigh, or upper arm). The dose will be reduced to 150 mg in the event of neutropenia, thrombocytopenia, and elevated liver enzymes.
  Interventions: Drug: Sarilumab 200 MG/1.14 ML Subcutaneous Solution [KEVZARA]

INTERVENTIONS:
Drug: Sarilumab 200 MG/1.14 ML Subcutaneous Solution [KEVZARA] — The treatment of sarilumab 200mg will be administered every two weeks subcutaneously.
  Each patient will be followed for 6 months from the start of treatment. The last administration of Sarilumab will be 2 weeks before the end of the study.

SUMMARY:
Rheumatoid arthritis (RA) is a condition associated with a high incidence of cardiovascular disease (CV), primarily as a result of accelerated atherosclerosis . Patients with RA also have a high prevalence of metabolic syndrome (MS) The state of chronic inflammation in RA patients contributes to increased CV risk.

Deregulation of both genetic and serological adipocines, MS biomarkers, and biomarkers of endothelial activation and inflammation also contributes to the increased CV risk in these patients.

An increased incidence of abnormal carotid intima-media thickness (cIMT) values and carotid plaques, considered surrogate markers of subclinical atherosclerotic disease, has also been described in patients with RA.

Positron emission tomography/computed tomography (PET/CT) is a noninvasive imaging technique useful for the evaluation of inflammation (by 18F-FDG uptake) and mineralization (by 18F-NaF uptake) in carotid atheroma plaque.

Atherosclerosis and RA share many common inflammatory pathways, and the mechanisms that lead to synovial inflammation are similar to those seen in atherosclerotic plaque.

Interleukin (IL)-6 is a key pro-inflammatory cytokine involved in both the pathophysiology of RA and the development of atherosclerosis.

Sarilumab is a human monoclonal antibody against the IL-6 receptor that has been shown to be effective in patients with RA, improving symptoms, as well as at the functional and radiographic levels.

Treatment with IL-6 receptor inhibitors has been described to result in a modulation of lipid metabolism, mediated by a reduction in lipoprotein (a) (Lp(a)) and an improvement in the anti-oxidant function of high-density lipoprotein (HDL) . In this regard, Sarilumab may have beneficial effects in RA patients on MS, which is implicated in the development of atherosclerotic disease.

Information regarding the beneficial effect of IL-6 receptor blockade on atheroma plaque formation and its effect at the vascular level in RA patients is scarce.

DETAILED DESCRIPTION:
RA is a chronic inflammatory disease characterized by chronic and erosive arthritis that mainly involves peripheral joints. RA affects activities of daily living, significantly decreasing the quality of life of affected patients. Several studies have demonstrated that RA patients are at higher risk of developing CV disease that is the main cause of premature mortality and sudden death in these patients. In this sense, the increased risk of CV disease observed in patients with RA is the result of a process of accelerated atherosclerosis. In addition, a large meta-analysis also found an increased prevalence of obesity, dyslipidemia, and hypertension, alterations in glucose metabolism and insulin resistance, which are features of MS, in patients with RA. Such characteristics are associated with inflammation and endothelial dysfunction, an early step of atherosclerosis. Besides traditional CV risk factors, the chronic inflammatory state present in these patients also contributes to the increased CV risk in RA. Moreover, CV risk in RA patients is further enhanced by a dysregulation both at the genetic and serological level of adipokines, MS-related biomarkers, biomarkers of endothelial activation and inflammation, which appear to be crucial in the development of atherosclerotic disease.

Accordingly, an adequate identification of patients at risk to develop CV events is needed. In this regard, carotid ultrasound and PET/CT are non-invasive techniques used to assess the extension and severity of atherosclerosis in RA. In this sense, molecular imaging techniques have the potential to study 'in vivo' the metabolic processes in the carotid atheroma. In fact, the incidence of abnormal cIMT values as well as the frequency of carotid plaques, which are surrogate markers of subclinical atherosclerotic disease, has been found increased in RA patients. In addition, it is well known that inflammation and mineralization are simultaneous phenomena in the atheroma plaque formation. In this regard, the uptake of 18F-FDG in relation with the inflammation of the carotid arteries has been demonstrated in patients with RA. Consequently, 18F-FDG may be considered as an established technique to evaluate the atheroma inflammation and to monitor the response to new anti-inflammatory therapies. Likewise, active calcification (which has a relevant role in the early phase of atherogenesis) measured by the uptake of 18F-NaF seems to be predominant over inflammation (18F-FDG) in symptomatic and asymptomatic carotid atheroma. This biological behavior opens new insights on the role of 18F-NaF in the study of calcification and in the identification of the vulnerable carotid atheroma.

Atherosclerosis and RA share many common inflammatory pathways, and the mechanisms leading to synovial inflammation are similar to those found in atherosclerotic plaque. Indeed, pro-inflammatory cytokines produced within locally affected joints in RA, such as IL-6, which regulates both the innate and adaptive immune system with a pivotal role in the pathophysiology of RA, are also central to the development of atherosclerosis. Specifically, IL-6 is a pleiotropic cytokine produced by a variety of cells types, including T-lymphocytes, macrophages, monocytes, endothelial cells and fibroblasts. This cytokine leads to the production of acute phase proteins in the liver, including serum CRP, among others. The production of IL-6 and thus CRP are key mediators of the systemic and local inflammation observed in RA. Furthermore, it is important to highlight that IL-6 has been shown to be significantly associated with atherosclerosis in RA patients. On the one hand, this molecule plays a direct role in mediating IR by inhibiting insulin receptor signal transduction and insulin action. On the other hand, IL-6 is independently predictive of endothelial dysfunction and a reduction in its serum levels leads to decreased endothelial cell activation in patients with RA. In addition, it has been demonstrated that the levels of Lp(a), a lipoprotein with atherogenic and thrombogenic properties, are higher in individuals with elevated IL-6 serum concentrations. Both IL-6 functions and its circulating levels are partially controlled by its receptor (IL-6R). Several studies have demonstrated a favourable effect on lipid metabolism with an anti-IL-6R treatment, besides reducing inflammatory disease activity. Moreover, a modulation of lipid metabolism, mediated by reduction of Lp(a) and improvement of the anti-oxidant role of HDL-cholesterol, has been reported in patients with RA following anti-IL-6R treatment. In this sense, Sarilumab (the first fully human anti-IL-6Rα monoclonal antibody) binds membrane-bound and soluble human IL-6R with high affinity, thereby blocking IL-6 signaling, with no evidence of complement-dependent or antibody dependent cell-mediated cytotoxicity. In preclinical studies, Sarilumab has been shown to inhibit IL-6 signaling in a dose-dependent manner. In phase II studies, SC Sarilumab was reasonably well tolerated and led to a decrease in acute-phase reactant levels, mainly in CRP in patients with RA. In addition, in RA patients treated with Sarilumab in combination with methotrexate, both drugs provided sustained clinical efficacy, significant improvements in symptomatic, functional, and radiographic outcomes are shown. In this regard, although it is plausible to think that the blockage of IL-6R may lead to a beneficial effect on atherosclerosis and MetS in patients with RA, this potential effect has not been extensively evaluated yet. With respect to this, little is known about the beneficial effect that IL-6R blockade may cause in the formation of atheroma plaque as well as the net vascular effect of lipids and lipoproteins changes in RA patients, which makes it a potent target of major interest.

Taking all these considerations into account, the aim of this study is to assess by PET/CT the effect of Sarilumab in the carotid atheroma plaque (effect on the inflammatory component as well as on mineralization) in patients diagnosed with RA over 6 months of Sarilumab treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years with active RA: DAS28>3.2 and PCR levels ≥1 mg/dL
2. Naïve to biological DMARDs or refractory to a single biological other than anti-IL-6 drugs.
3. Only patients with plaques detected by carotid ultrasound (at least 1.5 mm) should have a PET/CT scan.
4. Patients who are candidates for Sarilumab according to the summary of product characteristics
5. Patients who sign the informed consent form.

Exclusion Criteria:

1. Previous history of CV events.
2. History of diabetes or chronic renal failure.
3. Absolute neutrophil count <2 x109/L.
4. Platelet count <150 x 103/μL.
5. Elevated transaminases (ALT or AST > 1.5 x LSN).
6. Active infection, including localized infection.
7. That have contraindicated the administration of Sarilumab.
8. Patients who are participating in another clinical trial or research project.
9. Refusal to participate in the study and to sign the consent form.
10. Pregnant or nursing women, or women of childbearing age who are not using an effective method of contraception.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-04-30 (Estimated); Primary Completion 2020-10-30 (Estimated); Study Completion 2021-04-30 (Estimated)

PRIMARY OUTCOMES:
Effect of Sarilumab on carotid atheroma plaque (effect on the inflammatory component) using ultrasound in patients with RA | 6 months
Effect of Sarilumab on carotid atheroma plaque (effect on the mineralization) using ultrasound in patients with RA | 6 months

SECONDARY OUTCOMES:
Change in PET/CT 18F-FDG uptake in the aortic wall | 6 months
  (inflammatory component)
Change in PET/CT 18F-FNa uptake in the aortic wall | 6 months
  (mineralization)
Determine disease activity with DAS 28 index (Rheumatoid arthritis disease activity index) with 4 items corresponding to low (DAS28 = 2.43), medium (DAS28 = 4.05), high (DAS28 = 6.32) or very high (DAS28 = 8.40) activity. | 6 months
  Clinical improvement
Determine disease activity with CDAI index ( number of painful and swollen joints with 28 joints, the activity assessment by the patient and the physician on a scale from 0 to 10 and the PCR in mg/dl) | 6 months
  Clinical improvement
Determine disease activity | 6 months
  Clinical improvement in SDAI
Routine inflammatory parameters | 6 months
  Clinical improvement in C-reactive protein (CRP) levels
Change in the index of insulin resistance. | 6 months
Change in the index of insulin sensitivity. | 6 months
Modulation of the lipid profile using blood test | 6 months
Changes in mRNA expression by gene expression studies | 6 months
Changes in serum adipocine levels by ELISA/multiplex Serological studies | 6 months
Change in levels biomarker levels biomarkers associated with MS by ELISA/multiplex Serological studies | 6 months
  Retinol binding protein 4 (RBP4): μg/mL Ghrelin: μmol/L
Change in levels biomarkers of endothelial cell activation and inflammation. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Miguel Ángel González-Gay Mantecón, MDPhD, Principal Investigator — hospital universitario marques Valdecilla

IPD SHARING:
Plan to Share IPD: No